CLINICAL TRIAL: NCT01536067
Title: A Multicenter Phase II Study of Ofatumumab and Bortezomib (OB) in Previously Untreated Patients With Waldenstrom Macroglobulinemia
Brief Title: Ofatumumab and Bortezomib in Treating Patients With Previously Untreated Waldenstrom Macroglobulinemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding was withdrawn
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 205011; NCI-2011-03816 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-02-10; First posted 2012-02-20 (Estimated); Results first posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-05

CONDITIONS: Waldenström Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — ofatumumab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (monoclonal antibody therapy) (Experimental): INDUCTION PHASE: Patients receive ofatumumab IV on days 1, 8, and 15 and bortezomib SC on days 8 and 15. Beginning on course 2, patients receive ofatumumab IV on days 1 and 15 and bortezomib SC on days 1, 8, and 15. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Beginning 8 weeks after course 4 of induction phase, patients receive ofatumumab IV on day 1 and bortezomib SC on days 1, 8, and 15. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: ofatumumab; Drug: bortezomib; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: ofatumumab — Given IV
  Other Names: Arzerra; HuMax-CD20
Drug: bortezomib — Given SC
  Other Names: LDP 341; MLN341; VELCADE
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well giving ofatumumab together with bortezomib works in treating patients with previously untreated Waldenstrom macroglobulinemia. Monoclonal antibodies, such as ofatumumab and bortezomib, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving ofatumumab together with bortezomib may be a better way to block cancer growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine overall response rate (complete response [CR] + partial response [PR] + minor response [MR]) of ofatumumab in combination with bortezomib.

SECONDARY OBJECTIVES:

I. Determine complete remission (CR) rate, near (n)CR rate, very good partial response (VGPR) rate and PR rate per new criteria.

II. Determine 5 year progression free survival (PFS). III. Determine time to progression and duration of response of ofatumumab in conjunction with bortezomib.

IV. Determine safety of ofatumumab in combination with bortezomib. V. Conduct laboratory correlates.

OUTLINE:

INDUCTION PHASE: Patients receive ofatumumab intravenously (IV) on days 1, 8, and 15 and bortezomib subcutaneously (SC) on days 8 and 15. Beginning on course 2, patients receive ofatumumab IV on days 1 and 15 and bortezomib SC on days 1, 8, and 15. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Beginning 8 weeks after course 4 of induction phase, patients receive ofatumumab IV on day 1 and bortezomib SC on days 1, 8, and 15. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, and then every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Waldenstrom Macroglobulinemia and presence of cluster of differentiation (CD)20+ tumor cells as determined by immune-histochemistry or flow cytometric analysis in bone marrow or representative lymphoid tissue specimen; to be deemed eligible, patients must meet at least one of the following criteria:

  * Rising immunoglobulin (Ig)M
  * Hemoglobin =< 10 g/dL
  * Platelet count =< 100 x 10^9/L
  * Symptomatic or bulky lymphadenopathy or organomegaly
  * Systemic manifestations of Waldenstrom Macroglobulinemia (WM), such as hyperviscosity symptoms (patients with symptoms of hyperviscosity syndrome must be treated with plasmapheresis to control the syndrome prior to enrollment), neuropathy, amyloidosis, cryoglobulinemia, B-symptoms, or recurrent bleeding
* Must have a measurable disease as defined by the monoclonal IgM level of 1 g/dL on serum protein electrophoresis (SPEP); if the level of IgM on SPEP is less than 1 g/dL in patients who meet any criteria in inclusion criteria 2, then the IgM level obtained from nephelometric measurement may be used to justify this criterion
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of =< 2
* Have a life expectancy of >= 3 months
* Absolute neutrophil count >= 1.0 x 10^9/L unless the result of disease infiltration of bone marrow
* Platelet count >= 50 x 10^9/L unless the result of disease infiltration of bone marrow
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x the institutional upper limit of normal (ULN)
* Total bilirubin =< 3 mg/dL or 1.5 x institutional ULN, whichever is lower
* Serum creatinine =< 3 mg/dL
* Female patients are either post-menopausal or surgically sterilized otherwise they must agree to use acceptable contraceptive methods (e.g. double barrier) during treatment
* Male subjects, even if surgically sterilized (i.e., status post vasectomy) must agree to one of the following:

  * Practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug
  * Completely abstain from heterosexual intercourse
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent prior to receiving any study related procedure

Exclusion Criteria:

* Pregnant and nursing female patients
* Prior anti-neoplastic therapy for WM; the use of plasmapheresis to manage the symptoms of hyperviscosity and other IgM paraprotein mediated symptoms is allowed and does not disqualify a patient from the study; if a patient undergoes plasmapheresis within 8 weeks of starting the study treatment then the IgM level prior to plasmapheresis should be used for response assessment; neoplastic use of glucocorticoids is prohibited during the screening and treatment period; patients with active hyperviscosity symptoms should not be enrolled in this study unless the symptoms resolve after plasmapheresis
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive study drug
* Received an investigational agent within 30 days prior to enrollment
* Known human immunodeficiency virus (HIV) positive
* Positive serology for hepatitis B (HB) defined as a positive test for hepatitis B surface antigen (HBsAg); in addition, if HBsAg is negative and hepatitis B core antibody (HBcAb) is positive, regardless of hepatitis B surface antibody (HBsAb) status, a HB deoxyribonucleic acid test will be performed and if HB DNA is positive the patient will be excluded; if a patient is HBsAg negative, HBcAb positive, and HBsAb positive, indicating past but not active infection, the patient will be included on the study
* Positive serology for hepatitis C (HC) defined as a positive test for Hep C by enzyme immunoassays (EIA), in which case reflexively perform a HC recombinant immunoblot assay (RIBA) on the same sample to confirm the result
* Diagnosis of a malignant disorder other than WM within 3 years of the study enrollment with the exception of completely resected non-melanoma skin cancer and successfully treated in-situ cancer
* Uncontrolled infection
* Hypersensitivity to bortezomib, boron, or mannitol
* Grade 2 or greater peripheral neuropathy; since WM is known to cause peripheral neuropathy (PN), if, in investigator's judgement, a patient has Grade 2 PN related to WM, then he/she can be enrolled onto the study; under no circumstances patient with greater than Grade 2 PN can be enrolled
* Myocardial infarction within 6 months of enrollment; New York Heart Association (NYHA) Class III or more heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias; arrhythmias requiring active therapy other than chronic stable atrial fibrillation; if a patient has an implanted cardiac pacemaker and is otherwise well can be enrolled onto this study after demonstrating normal ejection fraction and clearance from a cardiologist; at the time of screening any electrocardiographic abnormality has to be documented as not medically relevant by the investigator before the patient proceeds to the enrollment phase
* Any serious medical or psychiatric illness that may interfere with participation in the study
* Patients with symptoms of hyperviscosity syndrome will not be enrolled on the study until they undergo plasmapheresis that results in resolution of symptoms and optimal control of the syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema Bhat, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Monoclonal Antibody Therapy): INDUCTION PHASE: Patients receive ofatumumab IV on days 1, 8, and 15 and bortezomib SC on days 8 and 15. Beginning on course 2, patients receive ofatumumab IV on days 1 and 15 and bortezomib SC on days 1, 8, and 15. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Beginning 8 weeks after course 4 of induction phase, patients receive ofatumumab IV on day 1 and bortezomib SC on days 1, 8, and 15. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  ofatumumab: Given IV
  bortezomib: Given SC
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Started | 3
Completed | 2
Not Completed | 1
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (CR + PR + MR) of Ofatumumab in Combination With Bortezomib
Description: Assessed using the Consensus Panel recommendations from the Third International Workshop on Waldenstrom Macroglobulinemia.
Time Frame: Every 28 days
Population: Due to the study's early termination and low accrual, data were not collected for this assessment.
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 0

2. Secondary Outcome: Frequency of Complete Remission (CR)
Time Frame: Every 28 days
Reporting Status: Not Posted

3. Secondary Outcome: Frequency of Near (n)CR
Time Frame: Every 28 days
Population: Due to the study's early termination and low accrual, data were not collected for this assessment.
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 0

4. Secondary Outcome: Frequency of Very Good Partial Response (VGPR)
Time Frame: Every 28 days
Population: Due to the study's early termination and low accrual, data were not collected for this assessment.
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Frequency of PR
Time Frame: Every 28 days
Population: Due to the study's early termination and low accrual, data were not collected for this assessment.
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Progression
Time Frame: From start of treatment to disease progression, assessed up to 12 months
Population: Due to the study's early termination and low accrual, data were not collected for this assessment.
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 0

7. Secondary Outcome: Progression-free Survival
Time Frame: From start of treatment to disease progression or death (regardless of the cause of death), whichever comes first, assessed up to 12 months
Population: Due to the study's early termination and low accrual, data were not collected for this assessment.
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 0

8. Secondary Outcome: Duration of Response
Time Frame: From the observation of a response to the time of disease progression, assessed up to 12 months
Population: Due to the study's early termination and low accrual, data were not collected for this assessment.
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 0

9. Secondary Outcome: Frequency and Severity of Toxicity as Graded According to the Cancer Therapeutic Evaluation Program (CTEP) Common Toxicity Criteria (CTC) Version 4.0
Description: Maximum grade per participant of any AE.
Time Frame: Every 30 days for 2 months
Population: All treated and eligible patients
Measure: Number; unit: participants
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Number analyzed (Participants) | 3
participants
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 3

ADVERSE EVENTS:
Arm/Group | Treatment (Monoclonal Antibody Therapy)
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Monoclonal Antibody Therapy) (N=3)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Iritis (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (2)
Gait disturbance (General disorders) | 1 (1)
Infusion site rash (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (1)
Injection site joint redness (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Furuncle (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (5)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Sensory loss (Nervous system disorders) | 1 (1)
Scrotal swelling (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Flushing (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes